CLINICAL TRIAL: NCT02472457
Title: Biologic and Immunomodulator Withdrawal in Pediatric Crohn Disease With Deep Clinical Remission Using the Crohn Disease Exclusion Diet
Brief Title: Crohn Disease Exclusion Diet After Single Medication De-escalation
Acronym: CEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-011628
Record Dates: First submitted 2015-06-10; First posted 2015-06-15 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Diet (Placebo Comparator): No dietary restrictions
  Interventions: Other: Free Diet
- Crohn Disease Exclusion Diet (Active Comparator): The CDED is a palatable diet that excludes foods suspected to have a role in intestinal inflammation.
  Interventions: Other: Crohn Disease Exclusion Diet

INTERVENTIONS:
Other: Crohn Disease Exclusion Diet — The CDED is divided into 4 stages: 0-6 weeks induction phase, weeks 7-12 step down phase, weeks 13-24 maintenance phase I, and weeks 25-52 maintenance phase II.
  Arms: Crohn Disease Exclusion Diet
Other: Free Diet — This diet contains no restrictions.
  Other Names: Placebo
  Arms: Free Diet

SUMMARY:
The primary objective of this study is to determine whether pediatric Crohn Disease (CD) patients in long-standing remission remain in remission longer after stopping medications if they follow the Crohn's Disease Exclusion Diet (CDED). The hypothesis is that subjects on the CDED will have longer time-to-relapse as opposed to those on an unrestricted diet.

DETAILED DESCRIPTION:
Crohn disease (CD) is an idiopathic, chronic, relapsing and remitting inflammatory condition of the gastrointestinal tract with a high risk for complications and need for surgical interventions, particularly in children. Immunomodulators and biologic therapies are effective at inducing and maintaining remission in pediatric CD, yet there is no proven strategy for reducing exposure to medications once sustained remission has been achieved. Diet has been proven to impact disease activity in CD and may allow for sustained drug-free remission. The primary objective of this study is to determine whether pediatric CD patients in long-standing remission remain in remission longer after stopping medications if they follow the Crohn's Disease Exclusion Diet (CDED). The hypothesis is that subjects on the CDED will have longer time-to-relapse as opposed to those on an unrestricted diet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Crohn Disease using the Revised Porto criteria who will be withdrawing from biologic or immunomodulator monotherapy as part of clinical care.
* Normal Growth Velocity, or Tanner 5
* Steroid-free Remission (Pediatric Crohn Disease Activity Index Score <10 without the height component) for at least 12 months prior to enrollment
* Colonoscopy during the preceding 3 months with complete mucosal healing or only few aphthous ulcerations located in one segment
* Stool calprotectin <250µg/g during the preceding 3 months
* Parental/guardian permission (informed consent) and, if appropriate, child assent.

Exclusion Criteria:

* Discontinuation of biologic or immunomodulator therapy by the subject without the approval of the primary gastroenterologist.
* Those subjects who in the judgment of the investigative team are unable to complete the study endpoints.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Stein, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Sigall-Boneh R, Pfeffer-Gik T, Segal I, Zangen T, Boaz M, Levine A. Partial enteral nutrition with a Crohn's disease exclusion diet is effective for induction of remission in children and young adults with Crohn's disease. Inflamm Bowel Dis. 2014 Aug;20(8):1353-60. doi: 10.1097/MIB.0000000000000110. PMID 24983973
- [Derived] Stein R, Daniel SG, Baldassano RN, Feigenbaum K, Kachelries K, Sigall-Boneh R, Weston S, Levine A, Bittinger K. Outcomes and Predictors of Sustained Remission After Drug Withdrawal in Pediatric Crohn Disease. J Pediatr Gastroenterol Nutr. 2022 Nov 1;75(5):608-615. doi: 10.1097/MPG.0000000000003589. Epub 2022 Aug 17. PMID 35976282

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Free Diet | Crohn Disease Exclusion Diet
Started | 8 (1 subject followed the Specific Carbohydrate Diet) | 11
Completed | 8 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Free Diet | Crohn Disease Exclusion Diet | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (3.6) | 16.0 (2.2) | 16.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
  Israel | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Sustained Relapse-free Remission
Description: Remission defined by the Pediatric Crohn Disease Activity Index, C-reactive protein, and stool calprotectin
Time Frame: At 52 weeks following enrollment
Population: 1 participant in the free diet group followed the specific carbohydrate diet and was in remission at 52 weeks. 1 participant in the CDED group withdrew prior to 52 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Free Diet | Crohn Disease Exclusion Diet
Number analyzed (Participants) | 8 | 9
Participants | 6 | 5

2. Secondary Outcome: Time-to-relapse
Description: Remission defined by the Pediatric Crohn Disease Activity Index, C-reactive protein, and stool calprotectin
Time Frame: Up to 104 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Microbial Composition of Gastrointestinal Tract (Types and Quantities of Microorganisms)
Description: Change in the microbial composition of the stool, mouth and rectum from baseline to 6 weeks
Time Frame: 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Microbial Composition of Gastrointestinal Tract (Types and Quantities of Microorganisms)
Description: Change in the microbial composition of the stool, mouth and rectum from baseline to 52 weeks
Time Frame: 52 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Dietary Compliance
Description: Using modified Medication Adherence Rating Scale (MARS) questionnaire
Time Frame: Up to 52 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Adverse event information was obtained via chart review and trial visits
Arm/Group | Free Diet | Crohn Disease Exclusion Diet
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT02472457/Prot_SAP_000.pdf